CLINICAL TRIAL: NCT06785376
Title: Estimating the Impact of a Multilevel, Multicomponent Intervention to Increase Uptake of HIV Testing and Biomedical HIV Prevention Among African-American/Black Gay, Bisexual and Same-gender Loving Men
Brief Title: P3 Trial: Estimating the Impact of a Multilevel, Multicomponent Intervention to Increase Uptake of HIV Testing and Biomedical HIV Prevention Among African-American/Black Gay, Bisexual, and Same-gender Loving Men
Acronym: P3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Victoria Anne Frye, Professor, Columbia University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: AAAU8754; R01MH129198 (NIH)
Record Dates: First submitted 2025-01-16; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: HIV Testing; PrEP Uptake
Keywords: HIV testing; PrEP uptake; HIV prevention; men who have sex with men
MeSH Terms: conditions — Homosexuality

STUDY DESIGN:
Intervention Model Description: A 2x2 factorial design to randomize and follow for 18 months 480 PrEP-eligible Black MSM (aged 18-65) living in the NYC area to one of four combinations: 1) SOC, DIY & TRUST; 2) SOC & TRUST (no DIY); 3) SOC & DIY (no TRUST); 4) SOC ALONE (no TRUST and no DIY). Hypotheses will be tested via regression (GEE) and Cox proportional hazard models; impact of the social/media campaign, delivered to both geographic (print media) and Black MSM communities (social media) and launched midway through recruitment, will be assessed through assessment of timing and length of exposure as covariates in the regression models and through interrupted time series methods.
Who Masked: Participant
Masking Description: We will endeavor to mask assignment with participants. It is possible (likely) that word will spread among networks of participants which arm is which. They of course are informed about the varying conditions/arms and that there are different numbers of sessions in each, but the exact "arm" is not disclosed to participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- A. SOC (Active Comparator): A. standard of care single-session, low threshold peer/near-peer navigation to PrEP.
  Interventions: Behavioral: SOC
- B. SOC & TRUST (Experimental): B. SOC standard of care single-session, low threshold peer/near-peer navigation to PrEP; TRUST single-session HIV self-testing training with facilitator
  Interventions: Behavioral: TRUST; Behavioral: SOC
- C. SOC & DIY (Experimental): C. SOC standard of care single-session, low threshold peer/near-peer navigation to PrEP; DIY three-session sexual health promotion/HIV prevention training with facilitator
  Interventions: Behavioral: DIY (Do It Yourself); Behavioral: SOC
- D. SOC, TRUST & DIY (Experimental): D. SOC standard of care single-session, low threshold peer/near-peer navigation to PrEP; TRUST single-session HIV self-testing training with facilitator; DIY three-session sexual health promotion/HIV prevention training with facilitator
  Interventions: Behavioral: DIY (Do It Yourself); Behavioral: TRUST; Behavioral: SOC

INTERVENTIONS:
Behavioral: DIY (Do It Yourself) — DIY is 3-session program that promotes empowerment, autonomy, stigma coping/resistance and social support to promote sexual health and pleasure and HIV prevention.
  Arms: C. SOC & DIY; D. SOC, TRUST & DIY
Behavioral: TRUST — TRUST is a single-session HIV self-testing training with facilitator
  Arms: B. SOC & TRUST; D. SOC, TRUST & DIY
Behavioral: SOC — standard of care single-session, low threshold peer/near-peer navigation to PrEP.

SUMMARY:
The major goal of this study is to evaluate a multi-component, multilevel HIV prevention intervention that targets theoretically-informed and empirically-identified barriers to and facilitators of both HIV testing and PEP/PrEP uptake by combining existing evidence-based and novel evidence-informed components and integrating them into a community-based organization's (CBO) standard of care (SOC) PEP/PrEP navigation program. The evaluation will apply use a 2x2 factorial design to randomize and follow for 18 months 480 PrEP-eligible Black MSM (aged 18-65) living in the NYC area to one of four combinations of interventions. The impact of the social/media campaign, delivered to both geographic (print media) and Black MSM communities (social media) and launched midway through recruitment, will be assessed through assessment of timing and length of exposure as covariates in analysis.

DETAILED DESCRIPTION:
The major goal of this study is to evaluate a multi-component, multilevel HIV prevention intervention that targets theoretically-informed and empirically-identified barriers to and facilitators of both HIV testing and PEP/PrEP uptake by combining existing evidence-based and novel evidence-informed components and integrating them into a community-based organization's (CBO) standard of care (SOC) PEP/PrEP navigation program. The existing evidence-based, individual-level component is TRUST (R01 DA-038108), a single-session peer-based HIV self-testing intervention for Black MSM. The existing, evidence-based community-level component is a social/print media campaign (CHHANGE [R21 MH-102182-01] & PEPTALK [R21 AI-122996]) to reduce community-level HIV stigma and drive demand for HIV testing, PEP and PrEP. The novel, evidence-informed, individual-level component is "Do It Yourself (DIY)", a 3-session enhancement of the CBO SOC peer navigation program that promotes empowerment, autonomy, stigma coping/resistance and social support via a novel "sexual self-care in-a-box" and peer-to-peer training to increase HIV testing and PEP/PrEP uptake.

The Specific Aims are:

1. Component test DIY, adapt social/print media campaign & manualize full intervention. We will conduct modified intervention mapping, component testing and post-test interviews with 20 PrEP-eligible Black MSM (for DIY) and focus groups with 20 PrEP-eligible Black MSM (for media campaign adaptation). A 15-person community consulting group of Black MSM, community leaders, media professionals, and service providers, will provide feedback on both components and the full manualized intervention.
2. Estimate main and interactive effects of components on recent HIV testing and PEP/PrEP uptake.

   H1: Exposure to TRUST, DIY, and the media campaign will each be associated with (1) higher past 3-month HIV testing; and (2) shorter time to PrEP uptake over time.

   H2: A multiplicative interaction among TRUST, DIY and length of exposure to the media campaign will emerge, such that exposure to combination of multiple interventions will be associated with the more positive outcomes compared to the impact of each intervention component individually.

   Primary outcomes: (1) HIV testing in past 3 months; (2) time to PrEP uptake: assessed via self-report, medical record, urine test (UrSure, qualitative, visually-read point of care test [validated machine analysis] measuring adherence to tenofovir, metabolite of tenofovir disopropil fumarate (TDF) and tenofovir alafenamide (TAF) via lateral flow immunoassay). Secondary outcomes:

   consistent HIV testing (2+ tests 3 months apart in 9 months), PEP uptake (self-report, medical record), PrEP/PEP adherence (self-report/ medical record/urine test). To test hypotheses, we will use a 2x2 factorial design to randomize and follow for 18 months 480 PrEP-eligible Black MSM (aged 18-65) living in NYC to one of four combinations: 1) SOC, DIY & TRUST; 2) SOC & TRUST (no DIY); 3) SOC & DIY (no TRUST); 4) SOC ALONE (no TRUST and no DIY). Hypotheses will be tested via regression (GEE) and Cox proportional hazard models; impact of the social/media campaign, delivered to both geographic (print media) and Black MSM communities (social media) and launched midway through recruitment, will be assessed through assessment of timing and length of exposure as covariates in the regression models and through interrupted time series methods.
3. Describe the feasibility, acceptability, and usability of intervention components and package via the Re-AIM implementation framework with an emphasis on component implementation by a CBO program.

ELIGIBILITY:
Inclusion Criteria:

1. assigned biological male sex at birth;
2. 18-65 years of age;
3. self-identify as: Black, African-American, Afro-Caribbean, Black African, Afro-Latino or multiethnic Black;
4. reside in the NYC metro area; (5) not HIV-positive (tested before randomization);

6) report insertive or receptive anal intercourse with another man in the past six months; 7) not currently on PEP or PrEP; 8) communicate in English or Spanish; 9) provide informed consent for the study.

Exclusion Criteria:

* Sexual identity is not an exclusion criterion
* potential participants who self-identify as Latino must also identify as Black (as per above) to be included

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
P3M HIV testing | past 3 months
  did the participant engage in HIV testing in the past 3 months
PrEP uptake | past 3 months
  PrEP uptake (yes/no)/time to PrEP uptake (assessed via self-report, medical record)

SECONDARY OUTCOMES:
consistent HIV testing | over 9 months
  consistent HIV testing (2+ tests 3 months apart in 9 months)
PEP uptake | past 3 months
  PEP uptake (self-report, medical record)
PrEP and PEP adherence | past 3 months
  PrEP/PEP adherence (self-report/medical record)

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided